CLINICAL TRIAL: NCT06292403
Title: Effect of Strength Training of Non-paretic Upper and Lower Limb With or Without Mirror Therapy on Motor Function Recovery of the Pareytic Side in Stroke Patients.
Brief Title: Effects of Strength Training of Non-paretic Upper and Lower Limb With or Without Mirror Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Farwa Akhtar
Record Dates: First submitted 2023-11-24; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Hemiplegic stroke; strength training AND stroke; Mirror therapy AND stroke; stroke rehabilitation; strength training and mirror therapy
MeSH Terms: conditions — Stroke | interventions — Resistance Training; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups
  1. Strength training only group
  2. strength training and mirror therapy group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training (Active Comparator): Non-hemiplegic lower limb stepping forward training Non-hemiplegic upper limb pulling elastic belt in standing position repeatedly Hemiplegic lower limb stepped over an obstacle or climbed a platform The patients will stretch their arms to touch distant objects in a standing position repeatedly.
  Interventions: Other: Strength Training
- Mirror Therapy and strength Training Group (Experimental): Participants in the (trial group) mirror and strength training group observed the reflection of the exercising arm and leg in the mirror. Participants in the (control group) strength training only group will exercise without a mirror entirely.
  Interventions: Other: Strength Training; Other: Mirror therapy

INTERVENTIONS:
Other: Strength Training — training time will be 30 minutes therapy, once a day, 3 days a week for 8 weeks. were allowed to rest for 3-5 min during each training.
Other: Mirror therapy — Participants in the (trial group) mirror and strength training group observed the reflection of the exercising arm and leg in the mirror. Participants in the (control group) strength training only group will exercise without a mirror entirely.
  Arms: Mirror Therapy and strength Training Group

SUMMARY:
The aim of this study is to find the effects of strength training with or without mirror therapy of non-paralytic upper limb for functional activities and in lower limb for gait pattern, balance and stability, and ADLs of paralytic side in patients with acute and sub-acute stroke. A randomized controlled trial that will include total 44 participants .The control group will undergo usual rehabilitation training along with strength training. The trial group will undergo strength training and mirror therapy of NHS on the basis of usual rehabilitation training. For the control group, training time will be 30 minutes, once a day, 3 days a week for 8 weeks. IN trial group, training time will be 30 minutes therapy, once a day, 3 days a week for 8 weeks. were allowed to rest for 3-5 min during each training. Data collected will be analyzed through SPSS 25.

DETAILED DESCRIPTION:
Stroke is defined as rapidly developing clinical signs of focal or global cerebral function disturbance that lasts more than 24 hours or leads to death, with no other apparent cause than that of vascular origin. Hemiplegia shows one side of the body paralysis involving one upper and one lower extremity. The term hemiplegia is often used generically to refer to the wide variety of motor problems that result from stroke.There are several stroke rehabilitation strategies for UL motor impairment including strength training and mirror therapy.

The idea is to re-educate the brain through a simple task, in which the individual performs a series of movements with the healthy arm, which is reflected in the mirror as if it was the injured arm. In this way, the reflex in the mirror of the healthy arm tricks the brain in believing that the injured arm is functioning as it should before the stroke. Isokinetic strengthening may provide motor and functional improvement in paretic upper extremity among patients with post-stroke hemiplegia. This strategy makes use of the brain's adaptability to enhance motor function after a stroke .

Monika Ehrensberger et al (2019) in a study concluded potential effectiveness of mirror-aided cross-education was undertaken and results portray that, in the case of training isometrically, cross-education was not augmented by mirror therapy. (The effectiveness of strength training of the NHS is evidenced in terms of promoting recovery in patients with stroke experiencing balance, mobility, and muscle strength of the paretic side .

Chenlan Shao et al (2022) conducted his study on the effect of strength training of the non-hemiplegic side (NHS) on balance function, mobility, and muscle strength of patients with stroke. He concluded that Strength training of the NHS can promote recovery of balance, mobility, and muscle strength of the paretic side of patients with stroke.

Harris et al demonstrated that leg weakness develops on the non hemiplegic side (NHS) in the first week after acute stroke. This decline in NHS muscle strength must not be ignored in patients with stroke, because it is highly associated with functional performance, and it can be used as an independent predictor of short-term functional gain and outcomes after stroke.

The previous study investigated the feasibility and potential effectiveness of mirror-aided cross-education compared with cross-education alone in post stroke upper limb recovery only. In addition, previous studies, mirror therapy, and contralateral strength training have shown promising results individually, but their direct comparison for both upper and lower limbs remains under-explored in the literature.

The rationale for this study stems from the critical need to understanding the effectiveness of only mirror-therapy performed solely versus mirror-aided treatment coupled with strength training in enhancing motor functionality across both upper and lower limbs can significantly impact rehabilitative protocols.

This research could uncover potential synergies between the two interventions, presenting an opportunity to develop cost effective novel combined approaches that capitalize on their respective strengths. Ultimately, the study's findings have the potential to advance the field of neuroplasticity aided neurorehabilitation and contribute to improved quality of life for individuals dealing with hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Girls aged 17-24 years with regular --Menstrual cycle
* Unmarried girls

Exclusion Criteria:

* Athletes
* Married women
* Girls who were regularly exercising
* Having any pelvic pathology
* Abnormal menstrual cycle.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Barthel Index | 8 weeks
  MBI is a five-level rating scale, including evaluation of bathing, grooming, feeding, dressing, bowels, bladder, toilet, stairs, chair/bed transfers, and walking. Higher scores represent higher degree of ADL independence. MBI was an efficient, reliable, and valid assessment of ADL for stroke patients.
Dynamic Gait Index | 8 weeks
  Dynamic Gait Index (DGI) is a performance-based tool that quantifies the dynamic balance instability developed by Shumway-Cook and Woollacott, evaluates the ability of the individual to modify gait in response to changing functions during walking.
Berg Balance Scale | 8 weks
  Consists of 14 tasks and total score of 56.score of 0-20 indicates severe fall risk, 20-45 includes moderate risk of fall and 45-60 illustrates thr functional balances state.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo Aabroo, Nmpt, Principal Investigator — Riphah International University
Locations (1):
- Fatima Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No